CLINICAL TRIAL: NCT00900016
Title: Pharmacodynamic Study of Fibroblast Activity Protein in Patients With Localized Pancreas Cancer Undergoing Surgical Resection
Brief Title: Studying Fibroblast Activity in Patients With Localized Pancreatic Cancer Undergoing Surgery
Status: Completed | Type: Observational
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000579635; 07-011 (Other: Fox Chase Cancer Center)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Pancreatic Cancer
Keywords: adenocarcinoma of the pancreas; recurrent pancreatic cancer; stage I pancreatic cancer; stage II pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Blotting, Western; Immunohistochemistry; Immunologic Techniques

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — peripheral blood sample
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: protein expression analysis
Genetic: western blotting
Other: immunohistochemistry staining method
Other: immunologic technique
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of tumor tissue and blood from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This research study is assessing fibroblast activity in patients with localized pancreatic cancer undergoing surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the degree of fibroblast activation protein (FAP) enzymatic activity at the tumor site in patients with localized pancreatic cancer.

Secondary

* To explore correlations between tumor stromal FAP enzymatic activity and stromal α_2-antiplasmin levels.
* To explore correlations between tumor FAP enzymatic activity and plasma dipeptidyl peptidase and plasma α_2-antiplasmin converting enzyme activity as potential surrogates.

OUTLINE: Patients undergo fine-needle aspiration of tumor or suspected mass at baseline. Tumor samples are analyzed by IHC for fibroblast activation protein (FAP) expression, immunocapture assay for ex vivo FAP enzymatic activity, and western analysis for FAP concentrations. Blood samples are collected weekly and analyzed for dipeptidyl peptidase activity by ELISA and α_2-antiplasmin converting enzyme.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Biopsy-proven adenocarcinoma of the pancreas or pancreatic mass suspicious for pancreatic cancer
* Localized disease
* Scheduled to undergo a resection or exploration of their pancreatic tumor

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Surgury patients scheduled to undergo a resection or exploration of their pancreatic tumor
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2007-08; Primary Completion 2013-12 (Actual); Study Completion 2017-06-23 (Actual)

PRIMARY OUTCOMES:
Independence of tumor fibroblast activation protein (FAP) activity and Met-α2-antiplasmin expression | Within 28 days for prior to surgery and at 3 month intervals for up to 2 years or recurrence

SECONDARY OUTCOMES:
Feasibility of exploiting the circulatory compartment to identify surrogates of tumor FAP | Within 28 days for prior to surgery and at 3 month intervals for up to 2 years or recurrence
Potential plasma surrogates of plasma dipeptidyl peptidase activity and plasma antiplasmin converting enzyme | Within 28 days for prior to surgery and at 3 month intervals for up to 2 years or recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Steven Cohen, MD, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania, United States